CLINICAL TRIAL: NCT02742376
Title: Comparison of Gait Parameters Between Floor and Sponge Surfaces and Special Shoes in Individuals With Difficulties in Weight-bearing
Brief Title: Comparison of Gait Parameters Between Floor and Sponge Surfaces and Special Shoes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Sponge- HMO-CTIL
Record Dates: First submitted 2016-03-02; First posted 2016-04-19 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-02

CONDITIONS: Arthroscopic Knee Surgery; Lower Limb Fractures; Back Pain and Asymmetric Gait; Complex Regional Pain Syndrome
MeSH Terms: conditions — Back Pain; Complex Regional Pain Syndromes | interventions — Floors and Floorcoverings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soft surface (Other): A soft sponge used for physiotherapy is placed on the floor along a path,
  Interventions: Other: Soft surface; Other: Floor; Other: Kyboot shoes
- Floor (Other): The subject will walk on the floor.
  Interventions: Other: Soft surface; Other: Floor; Other: Kyboot shoes
- Shoes (Other): Special shoes (Kyboot) with air cushions that are meant to relieve pressure will be used.
  Interventions: Other: Soft surface; Other: Floor; Other: Kyboot shoes

INTERVENTIONS:
Other: Soft surface — A sponge rectangle used in physiotherapy will be placed on the floor,
Other: Floor — A marked path on the floor where the subject is instructed to walk.
Other: Kyboot shoes — Special shoes will be worn by the subject.

SUMMARY:
This study compares the gait pattern of individuals with weight bearing difficulties walking on the floor, a soft surface, or with special shoes (Kyboot).

ELIGIBILITY:
Inclusion Criteria:

* 3 days to 1 month following arthroscopic knee surgery(n=10)
* Following fractures in lower limb with pain during weight-bearing (n=10)
* Back pain and asymmetrical gait (n=10)
* Complex Regional Pain Syndrome with pain during weight-bearing (n=10)

Exclusion Criteria:

* Neurological condition that does not permit walking on soft surface (drop foot)
* Wounds on feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Gait velocity | Two hours
  velocity [m/s]

SECONDARY OUTCOMES:
Step length | Two hours
  Step length [cm]
Base width | Two hours
  Base width [cm]
Cadence | Two hours
  Cadence [steps/s]
Single limb support duration | Two hours
  Single limb support time [s and % gait cycle time]
Double limb support duration | Two hours
  Double limb support time [s and % gait cycle time]